CLINICAL TRIAL: NCT01074619
Title: Effects of Memantine on Cognitive Disorders of Relapsing-remitting Multiple Sclerosis
Brief Title: Study on Cognitive Disorders of Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Ministry of Health, France (Other Government); H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-087
Record Dates: First submitted 2005-09-12; First posted 2010-02-24 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Memantine
  Interventions: Drug: Memantine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — 5 mg the first week, then 10 mg the second week, 15 mg the third week and finally 20 mg the fourth week until the end of the study (t0 + 1 year)
  Arms: 1
Drug: Placebo — 5 mg the first week, then 10 mg the second week, 15 mg the third week and finally 20 mg the fourth week until the end of the study (t0 + 1 year)
  Arms: 2

SUMMARY:
The purpose of this study is to determine if memantine is effective in the treatment on cognitive disorders of Relapsing - Remitting multiple sclerosis. m

ELIGIBILITY:
Inclusion Criteria:

* Remitting Multiple Sclerosis defined by Mc Donald et al., 2001
* Patient with authorised immunomodulator treatment or oral immunosuppressive therapy during more than three months: Bétâ Interferon, glatiramer acetate, azathioprine, methotrexate, mycophenolate mofetil, treatment by monoclonal antibody I.V. or anti-VLA4, natalizumab (Tysabri)
* Patient having benefited, possibly, of following treatments : mitoxantrone, cyclophosphamide, cyclosporine, general-purpose immunoglobulins, only if the treatment is ended more of 6 months before the inclusion.
* EDSS score ≤ 5.5
* DRS score ≥ 130
* PASAT 3s score > 15 and < median / control subjects according to 2 age brackets, sex, school level.
* Signed the informed consent form.
* Effective contraception for women in age to procreate

Exclusion Criteria:

* Progressive form MS
* MS relapse of less of 4 weeks.
* IV or oral corticoid treatment in the month preceding the screening
* Medicinal treatments or non medicinal in cognitive or psychology-stimulant aim in the 3 months before the screening
* Tumoral form MS visible in the MRI.
* Depressive syndrome (MADRS score > 19).
* Quite other diagnosed psychiatric pathology
* Known allergy or quite contraindication in memantin : renal or hepatic insufficiency, turned out epileptic disease, treatment by ketamine, amantadin, dextromethorphan, L-Dopa, dopaminergic agonist, barbituric, neuroleptic, 3,4-diaminopyridine, lithium, cimetidine, ranitidine, procainamide, quinine, nicotine, hydrochlorthiazide and ally, phenytoin, modafinil.
* Recent treatment (less of 4 weeks) by antidepressants and/or anxiolytics.
* Pregnancy or feeding.
* Minor or Major "protected by the law" patient
* Uncontrolled diet.
* Patient having benefited of one psychometric assessment(including in particular tests planned in the protocol) since less of one year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2005-09; Primary Completion 2011-03 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pace Auditory Serial Addition Test(P.A.S.A.T) | +1 year

CONTACTS AND LOCATIONS:
Overall Officials: Defer Gilles, Professor, Principal Investigator — Centre Hospitalier Universitaire de Caen
Locations (1):
- CHU Caen, Caen, France

REFERENCES:
- [Derived] Peyro Saint Paul L, Creveuil C, Heinzlef O, De Seze J, Vermersch P, Castelnovo G, Cabre P, Debouverie M, Brochet B, Dupuy B, Lebiez P, Sartori E, Clavelou P, Brassat D, Lebrun-Frenay C, Daplaud D, Pelletier J, Coman I, Hautecoeur P, Tourbah A, Defer G. Efficacy and safety profile of memantine in patients with cognitive impairment in multiple sclerosis: A randomized, placebo-controlled study. J Neurol Sci. 2016 Apr 15;363:69-76. doi: 10.1016/j.jns.2016.02.012. Epub 2016 Feb 6. PMID 27000224